CLINICAL TRIAL: NCT06400381
Title: Effectiveness of Mindfulness-Based Interventions on Professional Quality of Life, Work Engagement, and Sleep Quality Among Pediatric Nurses in Jordan
Brief Title: Effectiveness of Mindfulness-Based Interventions on Professional Quality of Life, Work Engagement, and Sleep Quality
Acronym: MBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20230532
Record Dates: First submitted 2024-04-16; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This study will be conducted using a 1-month prospective quasi-experimental design. The participants in this study are Jordanian pediatric nurses from different pediatric departments four major hospital in northern and central Jordan. Based on G power a satisfactory sample size for two groups (experimental group and control group) with a power level of 0.8, significant alpha level of 0.05, and a moderate effect size of 0.25 will be at least 80 participants for each group and 160 in total. To count for potential attrition, the investigators added additional 30% of the total sample to the participant resulting in a total sample size of 208 (104 in each group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Intervention (Experimental): There are many mindfulness-based interventions protocol that can be implemented and practice by healthcare organization. In the current study, the intervention protocol the investigators will use is based on Smiths version of mindfulness meditation (Smith, 2005). This version is compromised of several components includes being mindful of breathing, thought, sounds, taste, body scan, and sitting. The initial educational session by power point presentation will be given to the participant to explain the intervention rationale and procedure of mindfulness in daily life. In addition to giving opportunity for the participant to ask questions during the educational session.
  Interventions: Behavioral: Mindfulness
- Control (No Intervention): The control group will not receive any intervention and will continue with their usual routines and work schedules. The control group completes the pretest questionnaire at the same time as the interventional group completes it, the posttest will be after the interventional group has finished the mindfulness intervention 8 weeks. The intervention sessions used in the experimental group will be delivered to the control group at the end of study.

INTERVENTIONS:
Behavioral: Mindfulness — There are many mindfulness-based interventions protocol that can be implemented and practice by healthcare organization. In the current study, the intervention protocol the investigators will use is based on Smiths version of mindfulness meditation (Smith, 2005). This version is compromised of several components includes being mindful of breathing, thought, sounds, taste, body scan, and sitting. The initial educational session by power point presentation will be given to the participant to explain the intervention rationale and procedure of mindfulness in daily life. In addition to giving opportunity for the participant to ask questions during the educational session.
  Arms: Mindfulness-based Intervention

SUMMARY:
The aim of this study is to examine the impact of a mindfulness-based intervention on professional quality of life, work engagement, and sleep quality in pediatric and neonatal nurses. A quasi-experimental pretest-posttest design will be used to evaluate the effectiveness of the mindfulness-based intervention on professional quality of life, work engagement, and sleep quality among pediatric and neonatal nurses. Pediatric and neonatal nurses (number = 208) will be conducted at King Abdullah Hospital, Rahmah Hospital, Al-Basher Hospital, and Jordan University Hospital after getting the Institutional Review Board (IRB) approval from Jordan University of Science and Technology, in addition to the IRB from the Ministry of Health. The nurses will be allocated into two groups, one as an interventional group and one as a control group, and the participants will be asked to complete the pretest questionnaire (baseline pre-intervention) and then the post-test at the end of the intervention (8 weeks after baseline). Data will be collected using online questionnaires of the study variables and a demographic questionnaire for the participants. Data will be analyzed using the Statistical Package for the Social Sciences (version 26).

DETAILED DESCRIPTION:
The main goal of this study is to assess professional quality of life, work engagement, and sleep quality among nurses in a pediatric and neonatal unit in Jordan. A secondary aim was to examine the impact of a mindfulness-based intervention on nurses' professional quality of life, work engagement, and sleep quality in pediatric and neonatal nurses. Quasi-experimental pretest-posttest design with two groups will be used to achieve the primary study goal. Pretest-posttest quasi-experimental design, where the experimental group received the mindfulness intervention, and the control group received no intervention.

The study was conducted at four major hospitals in northern and central Jordan after getting IRB approval from the Jordan University of Science and Technology and research settings. The participants in this study Jordanian nurses were recruited from two different departments one is the Pediatric Intensive Care Unit (PICU) and the second department is Neonatal Intensive Care Unit (NICU).

The participants were invited to participate in the study through direct invitations by a member of the research team. The study was fully explained to them and informed consents were obtained from each individual participant. The nurses were assigned into two groups, one as an interventional group, and one as a control group. The intervention group who were willing to attend the mindfulness sessions participated in the intervention. The participants were invited to complete the data collection surveys to collect the baseline data. Then, the intervention group participants participated in the mindfulness-based intervention program. After completing the intervention, 8 weeks after baseline, post-intervention data were collected.

ELIGIBILITY:
Inclusion Criteria:

* Jordanian nurses
* nurses have at least one year experience in workplace setting

Exclusion Criteria:

* nurse manager
* staff have previous experience with any type of mindfulness-based intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Compassion fatigue | Change from baseline to 1-Month and 3 months post randomization
  The Professional Quality of Life Scale, version 5 which consisted of 30 items to assess nurses in three subscales: compassion satisfaction (CS), Burnout (BO), and secondary traumatic stress (STS), each subscale comprised 10 items. Nurses respond to each item of this questionnaire based on a 5-point Likert-type scale ranging from 1 (Never) to 5 (Very Often). The total scores range from 22 to 42 for each subscale. The first range of score is 22 or less indicates to lower scores, between 23-41 indicates moderate scores, and last range 42 or more indicates higher scores for each 3 subscales
Sleep Quality | Change from baseline to 1-Month and 3 months post randomization
  The Pittsburgh Sleep Quality Index (PSQI). The PSQI has 19 self-rated items grouped into seven components, these components are (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbance, (6) use of sleeping medication, and (7) daytime dysfunction. Scoring ranges from 0-3 points for each of the 7 components. The seven component scores are then summed to yield a global PSQI score, the global score ranges between 0 to 21. 0 indicates no difficulty on sleep and 21 indicates significant poor in sleep quality, and the global cutoff score of 5. Nurses with a score from 0 to 5 were regarded to have a good sleep quality, whereas nurses with a score of 6 to 21 or more than 5 were considered to have a poor sleep quality.
Work Engagement | Change from baseline to 1-Month and 3 months post randomization
  The Work Engagement Scale of Utrecht (UWES). The UWES consists of 17 items, and it includes three subscale of work engagement: Vigor (6 items), dedication (5 items), and absorption (6 items). Each item has a 7-point Likert response options ranging from 0 (Never) to 6 (Always). The total score for each subscale is calculated by summing the scores of the items in that dimension, the range of possible scores for each subscale is from 0 to 42. The total score for 17 items ranges from 0 to 102 with higher the scores indicating more nurses work engagement. For the sake of the current study, the investigators used the total score. The scores are classified as follows: very low (score < 5 percentile), low (5 percentile <= score < 25 percentile), average (25 percentile <= score < 75 percentile), high (75 percentile <= score < 95 percentile), and very high (95 percentile <= score).
Mindfulness | Change from baseline to 1-Month and 3 months post randomization
  The Five Facets of Mindfulness Questionnaire (FFMQ). The FFMQ consists of 39 items that measures five facets of mindfulness: Acting with Awareness (8 items e.g., I am easily distracted), Non-Judging of Experience (8 items e.g., I criticize myself for having irrational or inappropriate emotions), Observing (8 items e.g., I notice the smells and aromas of things), non-reactivity (7 items e.g., I watch my feelings without getting lost in them), and Describing (8 items e.g., I'm good at finding the words to describe my feelings). Each item was rated on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). The FFMQ scores is calculated by summing the scores on each item. The scores range from 8 to 40 (with the exception of the non-reactivity score which range from 7 to 35), with higher scores viewing greater mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al-Hammouri, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Alabdali Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared with other researchers. Only aggregate data will be disseminated.